CLINICAL TRIAL: NCT03790930
Title: Deep-learning Based Classification of Spine CT
Acronym: DETECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Shisheng He, MD, Executive Director of Orthopedic Department, Shanghai 10th People's Hospital
Other Study IDs: SHSY180624
Record Dates: First submitted 2018-11-16; First posted 2019-01-02 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Surgical Procedure, Unspecified
MeSH Terms: interventions — Deep Learning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- thin layer CT: Thin-layer CT will be manually labeled and used to train, validate and test deep learning algorithm.
  Interventions: Diagnostic Test: deep learning

INTERVENTIONS:
Diagnostic Test: deep learning — manually labeled samples will be used to train, validate and test deep learning algorithm, and then realize automatic classification.

SUMMARY:
It is time-consuming for spine surgeons or radiologists to conduct manual classifications of spinal CT, which may also be correlated with high inter-observer variance. With the development of computer science, deep learning has emerged as a promising technique to classify images from individual level to pixel level. The main of the study is to automatically identify and classify the lesions, or segment targeted structures on spinal CT with deep learning.

DETAILED DESCRIPTION:
Computer tomography (CT) is one of the most important imaging tool to assist the diagnostic and treatment of spinal disease. Classification of specific targets (e.g. individuals, lesions, etc.) is one of the most common mission of medical image analysis. However, it is time-consuming for spine surgeons or radiologists to conduct manual classifications of spinal CT, which may also be correlated with high inter-observer variance. With the development of computer science, deep learning has emerged as a promising technique to classify images from individual level to pixel level. The main of the study is to automatically identify and classify the lesions, or segment targeted structures on spinal CT with deep learning.

ELIGIBILITY:
Inclusion Criteria:

- spinal thin layer CT

Exclusion Critera:

* medals or other implants induce artifact
* poor image quality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with thin layer spinal CT covering targeted level will be included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
classification accuracy | 1 day
  classification accuracy (e.g. area under the curve, etc.)
segmentation accuracy | 1 day
  segmentation accuracy of multiple structures (e.g. Dice score, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Shisheng He, M.D., Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided